CLINICAL TRIAL: NCT05797610
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Sefaxersen, an Antisense Inhibitor of Complement Factor B, in Patients With Primary IgA Nephropathy at High Risk of Progression
Brief Title: A Study to Evaluate the Efficacy and Safety of Sefaxersen (RO7434656) in Participants With Primary Immunoglobulin A (IgA) Nephropathy at High Risk of Progression
Acronym: IMAGINATION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WA43966; 2022-502102-32-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sefaxersen (RO7434656) (Experimental): Participants will receive subcutaneous (SC) doses of sefaxersen (RO7434656) on Days 1, 15, and 29 followed by once every 4 weeks (Q4W) until Week 105. Participants may be eligible to switch to open-label treatment after Week 105 at the investigator's discretion until up to 1 year after the common-close timepoint, the date when the last participant completes the Week 105 assessment, withdraws, or is discontinued from the study.
  Interventions: Drug: Sefaxersen (RO7434656)
- Placebo (Placebo Comparator): Participants will receive SC doses of sefaxersen (RO7434656) matching placebo on Days 1, 15, and 29 followed by once Q4W until Week 105. Participants may be eligible to switch to open-label treatment after Week 105 at the investigator's discretion until up to 1 year after the common-close timepoint, the date when the last participant completes the Week 105 assessment, withdraws, or is discontinued from the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sefaxersen (RO7434656) — Sefaxersen (RO7434656) will be administered as SC injection per schedule as specified.
  Other Names: Sefaxersen
  Arms: Sefaxersen (RO7434656)
Drug: Placebo — Matching placebo will be administered as SC injection per schedule as specified.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of sefaxersen (RO7434656), a novel Antisense Oligonucleotide (ASO) therapy in participants with primary IgA nephropathy (IgAN) who are at high risk of progressive kidney disease despite optimized supportive care.

ELIGIBILITY:
Inclusion Criteria:

* Primary IgAN, as evidenced by a kidney biopsy performed within 10 years prior to or during screening, without known secondary cause
* Treatment with maximum tolerated doses of angiotensin-converting enzyme (ACE) inhibitors or angiotensin II receptor blockers (ARBs) for at least 90 days immediately prior to screening, and without an intent to modify the dose during the study, except for interruptions due to illness (not greater than 7 consecutive days), unless the potential participant is intolerant to these medications
* Urine Protein-to-Creatinine Ratio (UPCR) ≥ 1 gram per gram (g/g) or urine protein excretion ≥ 1 gram per day (g/day) (with UPCR ≥ 0.8 g/g), all measured from a 24-hour urine collection during screening
* eGFR ≥ 20 mL/min/1.73 m^2, as calculated by the 2021 CKD-EPI creatinine equation (Inker et al. 2021a)
* Vaccination against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae according to national vaccination recommendations
* Female participants of childbearing potential must use adequate contraception

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 12 weeks after the final dose of sefaxersen
* Histopathologic or other evidence of another autoimmune glomerular disease
* Presence of ≥ 50% crescents on kidney biopsy, sustained doubling of serum creatinine within 3 months prior to screening, or rapidly progressive glomerulonephritis in the opinion of the investigator
* History of kidney transplantation
* Glycated Hemoglobin (HbA1c) ≥ 6.5% or a clinical diagnosis of diabetes mellitus of any type
* Systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg from the average of two measurements performed at least 1 minute apart during screening
* Initiation of sodium-glucose cotransporter-2 (SGLT2) inhibitors within 16 weeks prior to screening or during screening
* Initiation of endothelin receptor antagonists within 90 days prior to screening or during screening
* Initiation of mineralocorticoid receptor antagonists or non-dihydropyridine calcium channel blockers within 90 days prior to screening or during screening
* Use of herbal therapies within 90 days prior to or during screening
* Treatment with investigational therapy within 28 days prior to screening or 5.5 drug-elimination half-lives of that investigational product prior to screening
* Treatment with an investigational therapy planned during the treatment period
* Previous treatment with sefaxersen
* Treatment with oral or intravenous (IV) corticosteroids with a dose equivalent to ≥ 7.5 milligrams per day (mg/day) of prednisone for 7 days or equivalent to ≥ 5 mg/day of prednisone for 14 days within 90 days prior to screening
* Treatment with corticosteroids with systemic effects during screening
* Treatment with a systemic calcineurin inhibitor within 2 months prior to screening or during screening
* Treatment with anti-CD20 therapy within 9 months of screening or during screening
* Treatment with other systemic immunosuppressive agents within 6 months of randomization including, but not limited to, complement inhibitors, alkylating agents (e.g., cyclophosphamide or chlorambucil), azathioprine, or mycophenolate
* Planned major procedure or major surgery during screening or the study
* Substance abuse within 12 months prior to screening or during screening
* Any serious medical condition or abnormality in clinical laboratory tests that precludes an individual's safe participation in and completion of the study
* History of malignancy within < 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Usage of Glucagon-like Peptide-1 (GLP-1)-based therapy (i.e., GLP-1 mono-agonists, GLP-1/GIP dual agonists, etc.) within 90 days prior to screening or during screening, or intent to initiate during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Urine Protein-to-Creatinine Ratio (UPCR) at Week 37 | Baseline, Week 37
  UPCR will be assessed in urine sampled over 24 hours.

SECONDARY OUTCOMES:
Estimated Glomerular Filtration Rate (eGFR) Slope at Week 105 from Baseline | Baseline, Week 105
  eGFR will be calculated using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation.
Time to the Composite Kidney Failure Endpoint | Up to approximately 36 months
  Time to the composite kidney failure endpoint is defined as receipt of kidney transplantation, need for kidney replacement therapy, or a sustained decline in eGFR of ≥ 30% or a sustained eGFR < 15 milliliters/minutes/1.73m^2 (mL/min/1.73m^ 2) over at least 4 weeks (both eGFR criteria requires two consecutive central laboratory eGFR values meeting criteria ≥ 4 weeks apart), whichever occurs first, without the receipt of other immunosuppressive or background therapies for the treatment of IgAN.
Change From Baseline in Fatigue at Week 105 | Baseline, Week 105
  Fatigue will be assessed with the Functional Assessment of Chronic Illness Therapy-Fatigue subscale (FACIT-F). The FACIT-F Scale is a 13-item scale used to measure self-reported fatigue. Items are assessed on a 5-point Likert scale, with responses ranging from 0 for "not at all" to 4 for "very much". The total raw score is the sum of the values of each scored question and ranges from 0 to 52. A higher score indicates less fatigue.
Percentage of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to approximately 36 months
Plasma Concentration of Sefaxersen | Up to approximately 36 months

OTHER OUTCOMES:
Change From Baseline in Symptoms and Health-Related Quality of Life at Week 105 as Assessed Using the RAND Kidney Disease and Quality of Life 36-Item (KDQOL-36) Short Form | Baseline, Week 105
  The RAND KDQOL-36 is an abbreviated questionnaire that combines the generic and disease-specific components to assess participant's health-related quality of life. This 36-item questionnaire includes the RAND 12, Version 1 (12 items) and 3 disease-related domains, symptoms/problems (12 items), burden of kidney disease (4 items), and effects of kidney disease (8 items). It uses a recall of 4 weeks, and items are assessed on 3- to 5-point Likert scales or with a dichotomous response option. Higher score indicates better health. The raw scores are transformed linearly to a range of 0 to 100, with higher scores indicating better health.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (198):
- United States (37):
  - Alabama Kidney Research - ERN - PPDS, Alabaster, Alabama
  - UAB Nephrology Research Clinic, Birmingham, Alabama
  - Sunrise Medical Management LLC, Surprise, Arizona
  - Tucson Neuroscience Research - M3 WR, Tucson, Arizona
  - Kidney Disease Medical Group Inc-1505 Wilson Ter, Glendale, California
  - Southern California Medical Research Center, La Palma, California
  - Academic Medical Research Institute - Los Angeles, Los Angeles, California
  - University of California, Los Angeles (UCLA) - Hematology/Oncology Santa Monica, Los Angeles, California
  - Los Angeles County Nephrology, Montebello, California
  - North America Research Institute-San Dimas, San Dimas, California
  - Hope Clinic & Research Center, Hialeah, Florida
  - LCC Medical Research - Miami - ClinEdge - PPDS, Miami, Florida
  - Central Florida Kidney Specialists, Orlando, Florida
  - L&C Professional Medical Research Institute, West Miami, Florida
  - Cowry Medical Group LLC, Acworth, Georgia
  - Care Institute Idaho Kidney Institute, Chubbuck, Idaho
  - Care Institute Idaho Kidney Institute, Idaho Falls, Idaho
  - Nephrology Associates of Northern Illinois, Hinsdale, Illinois
  - University of Iowa, Iowa City, Iowa
  - Massachussets General Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Sierra Nevada Nephrology Consultants, Reno, Nevada
  - NYU Langone Nephrology Associates - Mineola, Mineola, New York
  - North Carolina Nephrology, PA, Raleigh, North Carolina
  - Ohio State University Wexner Medical Center - Outpatient Care East, Columbus, Ohio
  - Kidney and Hypertension Center, Roseburg, Oregon
  - Austin Diagnostic Clinic - Frenova F1, Austin, Texas
  - Global Medical Research - M3 WR, Dallas, Texas
  - Texas Kidney Institute - Dallas, Dallas, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - R & H Clinical Research, Katy, Texas
  - Revival Research Corporation - Sherman - ClinEdge - PPDS, Sherman, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - Nephrology Associates of Northern Virginia Inc, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Milwaukee Nephrologists, Sc, Wauwatosa, Wisconsin
- Argentina (5):
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Ciudad Autonoma Buenos Aires
  - Consultorios Médicos Dr. Doreski, Ciudad Autonoma Buenos Aires
  - Sanatorio Mayo Privado, Córdoba
  - Sanatorio Allende, Córdoba
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
- Australia (7):
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Brazil (7):
  - Santa Casa de Misericordia de Belo Horizonte - PPDS, Belo Horizonte, Minas Gerais
  - Freire Pesquisa Clinica, Belo Horizonte, Minas Gerais
  - Hospital de Clinicas de Porto Alegre HCPA PPDS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clinica da Fundação Pró Rim, Joinville, Santa Catarina
  - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Hospital Do Rim E Hipertensao Fundacao Oswaldo Ramos, São Paulo, São Paulo
  - Instituto D?Or Pesquisa e Ensino - Hospital Gloria D?Or, Rio de Janeiro
- Canada (6):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Cape Breton Regional Hospital, Sydney, Nova Scotia
  - London Health Sciences Centre · Victoria Hospital, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- China (25):
  - Beijing Friendship Hospital, Capital Medical University - PPDS, Beijing, Beijing Municipality
  - Cangzhou Central Hospital, Cangzhou Shi, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Changzhou First People's Hospital, Changzhou
  - West China Hospital, Sichuan University, Chengdu
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhejiang Provincial People?s Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Ningbo No.2 Hospital, Ningbo
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Xinhua Hospital Affiliated To Shanghai Jiaotong University School of Medicine, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (6):
  - Centre Hospitalier, Annonay
  - CHU Boulogne sur Mer, Boulogne-sur-Mer
  - Hopital Henri Mondor, Créteil
  - Hopital Tenon, Paris
  - Hopital Bichat - Claude Bernard AP-HP, Paris
  - Hôpital de Rangueil, Toulouse
- Germany (6):
  - Universitatsklinikum der RWTH Aachen, Aachen
  - St. Joseph-Krankenhaus, Berlin
  - Klinikum Koln-Merheim, Cologne
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen
- Greece (4):
  - University General Hospital of Heraklion, Heraklion
  - Venizeleio General Hospital of Heraklion, Heraklion
  - University General Hospital of Patras, Pátrai
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Queen Mary Hospital, Hong Kong, Hong Kong
- Italy (7):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, Apulia
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi-Via Massarenti, Bologna, Emilia-Romagna
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Ospedale Policlinico San Martino, Genoa, Liguria
  - IRCCS Pavia - Istituti Clinici Scientifici Maugeri Spa ? Società Benefit, Pavia, Lombardy
  - Ospedale San Giovanni Bosco, Turin, Piedmont
- Japan (30):
  - Fujita Health University Hospital, Aichi
  - Hirosaki University Hospital, Aomori
  - Juntendo University Urayasu Hospital, Chiba
  - University of Yamanashi Hospital, Chūō
  - Matsuyama Red Cross Hospital, Ehime
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Hokkaido University Hospital, Hokkaido
  - Tokyo Medical University Ibaraki Medical Center, Inashiki-Gun
  - Kanazawa Medical University Hospital, Ishikawa
  - Nara Medical University Hospital, Kashihara
  - Kumamoto University Hospital, Kumamoto
  - Tohoku University Hospital, Miyagi
  - Kyoto City Hospital, Nakagyo-ku
  - Nara Prefecture General Medical Center, Nara
  - Hyogo Prefectural Nishinomiya Hospital, Nishinomiya
  - Iwate Medical University Hospital, Numakunai
  - National Hospital Organization Okayama Medical Center, Okayama
  - Okayama University Hospital, Okayama-Shi Kita-Ku
  - University of the Ryukyus Hospital, Okinawa
  - Saitama Medical University Hospital, Saitama
  - Osaka University Hospital, Suita
  - Jichi Medical University Hospital, Tochigi
  - Tokushima University Hospital, Tokushima
  - The Jikei University Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Juntendo University Nerima Hospital, department of renal and hypertension, Tokyo
  - University of Tsukuba Hospital, Tsukuba
  - Yamaguchi University Hospital, Ube
- Malaysia (8):
  - Hospital Kuala Lumpur, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Seri Manjung, Seri Manjong, Pahang
  - Taiping Hospital, Taiping, Perak
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Ampang, Ampang
  - Miri Hospital, Miri
- Mexico (5):
  - Clinica San Cosme, Fracc Lomas Del Campestre, Aguascalientes
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Barrio Belisario Domínguez Secc XVI, Mexico CITY (federal District)
  - Centro de Investigacion Clinica Chapultepec S. A. de C. V., Morelia, Michoacán
  - Instituto Mexicano de Trasplantes, Cuernavaca, Morelos
  - Christus Latam Hub Center Of Excellence & Innovation, Monterrey, Nuevo León
- Poland (7):
  - 4. Wojskowy Szpital Kliniczny z Poliklinika SP ZOZ, Wroclaw, Lower Silesian Voivodeship
  - SCM Clinic - Prywatny Szpital Specjalistyczny, Krakow
  - SPZOZ Centralny Szpital Klin, Lodz
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Szpital Kliniczny im. H.Swiecickiego UM w Poznaniu, Późna
  - Szpital Kliniczny Dzieciatka Jezus, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroc?aw
- Singapore (4):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
- South Korea (11):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Chungbuk National University Hospital, Cheongju-si
  - Ajou University Hospital, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Gangdong Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Spain (7):
  - Hospital Universitari Arnau de Vilanova, Lleida, Lerida
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Ribera Polusa, Lugo
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Medical Foundation, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Far Eastern Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
  - Taichung Veterans General Hospital, Xitun Dist.
  - Mackay Memorial Hospital-Taipei branch, Zhongshan Dist.
- United Kingdom (6):
  - Addenbrookes Hospital, Cambridge
  - Leicester General Hospital, Leicester
  - Guys and St Thomas Hospital, London
  - Kings College Hospital, London
  - Churchill Hospital, Oxford
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Tekendo-Ngongang C, Gleeson JG, Mignon L. Treating the Untreatable: Antisense Oligonucleotides as an Individualized Therapy for Rare Genetic Kidney Diseases. J Am Soc Nephrol. 2024 Dec 1;35(12):1774-1777. doi: 10.1681/ASN.0000000532. Epub 2024 Sep 27. No abstract available. PMID 39331470
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639